CLINICAL TRIAL: NCT04617236
Title: Cultivando la Salud: A Breast and Cervical Cancer Screening Promotion Program for Low-Income Puerto Rican Women
Acronym: CLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Vivian Colon, Professor, University of Puerto Rico
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: A1250312
Record Dates: First submitted 2020-10-14; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: Hispanic women; Behavioral Intervention; Lay Health Workers
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial using a pre-post comparison group design. Eligibility criteria included ages 21 and older for the Pap cohort and 40 and older for the mammography cohort, non-adherence to recommended Pap test screening and/or mammography screening guidelines according to the American Cancer Society, no hysterectomy, no diagnosis of cancer, and not currently pregnant. Trained data collectors administered a baseline survey to eligible women and randomly assigned them to the intervention or to a comparison condition. Lay Health Workers delivered the intervention in women's homes, and administered the follow-up survey by phone 4 to 6 months following baseline.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cultivando la Salud Educational Intervention (Experimental): After completing eligibility and baseline surveys, Lay health workers delivered an educational intervention for breast and cervical cancer screening. This educational session was delivered in participants' home and lasted between 1-2 hours. Follow-up data was collected 4-6 months post educational session.
  Interventions: Behavioral: Cultivando La Salud
- Control (No Intervention): No intervention was delivered. At baseline, participants completed eligibility and baseline surveys. Follow-up data was collected 4-6 months post-baseline survey.

INTERVENTIONS:
Behavioral: Cultivando La Salud — A lay health worker delivered educational intervention for breast and cervical cancer screening.
  In total, the Intervention Group subject participation will take approx. up to four hours (1 hour for interview, 1 hour for the second interview, and 1-2 hours for the CLS intervention) and Control Group up to four hours (One hour for interview, one hour for the second interview, up to two hours for educational intervention after the second interview).
  Follow-up data was collected 4-6 months post education session (intervention group) or post-baseline survey (control group).
  Arms: Cultivando la Salud Educational Intervention

SUMMARY:
The overall goal of this education program is to increase breast and cervical cancer screening in low-income women in Puerto Rico through implementation of an evidence-based educational program that addresses both health professionals (promotoras or community health workers) and public audiences of low-income women living in Canóvanas, Puerto Rico who have either never been screened for breast and/or cervical cancer, or are under-screened according recommended guidelines. To evaluate promotoras' delivery of the CLS screening education program we used a randomized pre-post comparison group study design that will provide data to determine the effectiveness of the CLS intervention program compared with usual practice (no intervention).

DETAILED DESCRIPTION:
The proposed promotora and community based breast and cervical screening education program includes the following specific aims:

Aim 1. To train community health workers (promotoras) from Taller Salud to implement the CLS breast and cervical cancer screening program. Taller Salud staff train and build capacity of promotoras to implement the CLS community-based education and navigation program.

Aim 2. To deliver the CLS intervention program to at least 600 women in Canóvanas municipality, Puerto Rico.

Aim 3. To evaluate the impact of the program on increasing mammography and cervical cancer screening among participating women in Canóvanas, Puerto Rico.

Aim 4. To adapt and update intervention materials

ELIGIBILITY:
Inclusion Criteria:

* Women aged 21 and older for Pap cohort
* Women aged 40 and older for Mammography cohort

Exclusion Criteria:

* Having completed a Papanicolau test in the past 3 years if participant is between the ages of 21-65.
* Having completed a Mammography screening in the past year if participant is aged 40 or older
* Have a hysterectomy
* Currently pregnant
* History of any type of cancer

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2012-05-15 (Actual); Primary Completion 2013-09-20 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Number of participants aged 21 and older who completed a cervical cancer screening (Pap test) | 4-6 months after the intervention
  Screening behavior status at baseline and follow-up were assessed by asking women the month and year of their last Pap test.
Number of participants aged 40 and older who completed a mammography test | 4-6 months after the intervention
  Screening behavior status at baseline and follow-up were assessed by asking women the month and year of their last mammogram.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Colón-López, PhD, Principal Investigator — Graduate School of Public Health, University of Puerto Rico Medical Sciences Campus
Locations (1):
- University of Puerto Rico, Medical Sciences Campus, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Colon-Lopez V, Gonzalez D, Velez C, Fernandez-Espada N, Feldman-Soler A, Ayala-Escobar K, Ayala-Marin AM, Soto-Salgado M, Calo WA, Pattatucci-Aragon A, Rivera-Diaz M, Fernandez ME. Community-Academic Partnership to Implement a Breast and Cervical Cancer Screening Education Program in Puerto Rico. P R Health Sci J. 2017 Dec;36(4):191-197. PMID 29220062